CLINICAL TRIAL: NCT00353483
Title: Effect of Neoadjuvant or Adjuvant Systemic Therapy on Breast Cancers, Bone Marrow Cancer Cells, and Circulating Cancer Cells
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 05-0648 / 201101961
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast cancer tissue, peripheral blood, and bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tissue, blood, and bone marrow (optional) collection: * Undergo neoadjuvant systemic therapy
    * initial surgery for sentinel lymph node biopsy/portacath placement
    * definitive cancer surgery (if applicable)
    * when portacath is removed (1 year, if available)
    * if metastatic disease develops or is present in accessible sites, a sample may be collected at the time of specimen collection for diagnosis
  * Undergo Adjuvant Systemic Therapy
    * initial surgery for a sentinel lymph node biopsy/portacath placement
    * when portacath is removed (1 year, if available)
    * If metastatic disease develops or is present in accessible sites, a sample may be collected at the time of specimen collection for diagnosis.
  * Undergone neoadjuvant systemic therapy
    * during definitive cancer surgery/portacath removal (if available)
    * if metastatic disease develops or is present in accessible sites, a sample may be collected at the time of specimen collection for diagnosis
  Interventions: Procedure: Peripheral blood draw; Procedure: Breast tissue collection; Procedure: Bone marrow biopsy

INTERVENTIONS:
Procedure: Peripheral blood draw
Procedure: Breast tissue collection
Procedure: Bone marrow biopsy

SUMMARY:
The main purpose of this study is to compare genetic markers present on tumor cells before and after chemotherapy.

DETAILED DESCRIPTION:
In this study, the investigators propose that persistent disseminated tumor cells (DTC) present after systemic therapy represent a unique subpopulation of all DTC, are predictors of a poor response to systemic therapy and correlate with poor clinical outcome. The investigators hypothesize that systemic therapy-resistant DTC can be identified by their expression of a unique constellation of tumor marker proteins which may be similar to those expressed by breast cancer stem cells. In this research, the investigators' specific aims are : 1) to characterize tumor markers expressed by DTC which are present after systemic therapy, 2) to compare the expression of these markers to that on DTC detected prior to systemic therapy, 3) to correlate expression of the defined tumor markers on DTC with clinical outcome of breast cancer patients to identify those markers that are predictive of disease recurrence, 4) to utilize biomarkers identified in Specific Aims 1 and 2 to isolate purified DTC for further molecular analysis.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed with clinical stage II, III, or IV breast cancer
* Planning to undergo neoadjuvant or adjuvant systemic therapy; patients who have already completed neoadjuvant systemic therapy are also eligible
* Must be >= 18 years of age
* If female, must not be pregnant
* Must not have Hepatitis B, C, or HIV
* Must be willing and able to sign informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in clinic at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2005-09-14 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Characterize tumor markers expressed by DTC which are present after systemic therapy | Approximately 6 years
Compare the expression of these markers to that on DTC detected prior to systemic therapy | Approximately 6 years
Correlate expression of the defined tumor markers on DTC with clinical outcome of breast cancer patients to identify those markers that are predictive of disease recurrence. | Approximately 6 years
Compare the tumor markers present on DTC before and after chemotherapy with the tumor marker expression of the primary tumor and post-treatment tumor. | Approximately 6 years.
To xenograft tumor cells into mice for further genetic and phenotypic characterization. | Approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Aft, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diel IJ, Cote RJ. Bone marrow and lymph node assessment for minimal residual disease in patients with breast cancer. Cancer Treat Rev. 2000 Feb;26(1):53-65. doi: 10.1053/ctrv.1999.0150. PMID 10660491
- [Background] Braun S, Pantel K, Muller P, Janni W, Hepp F, Kentenich CR, Gastroph S, Wischnik A, Dimpfl T, Kindermann G, Riethmuller G, Schlimok G. Cytokeratin-positive cells in the bone marrow and survival of patients with stage I, II, or III breast cancer. N Engl J Med. 2000 Feb 24;342(8):525-33. doi: 10.1056/NEJM200002243420801. PMID 10684910
- [Background] Braun S, Naume B. Circulating and disseminated tumor cells. J Clin Oncol. 2005 Mar 10;23(8):1623-6. doi: 10.1200/JCO.2005.10.073. No abstract available. PMID 15755968
- [Background] Janni W, Rack B, Schindlbeck C, Strobl B, Rjosk D, Braun S, Sommer H, Pantel K, Gerber B, Friese K. The persistence of isolated tumor cells in bone marrow from patients with breast carcinoma predicts an increased risk for recurrence. Cancer. 2005 Mar 1;103(5):884-91. doi: 10.1002/cncr.20834. PMID 15666325
- [Background] Klein CA, Blankenstein TJ, Schmidt-Kittler O, Petronio M, Polzer B, Stoecklein NH, Riethmuller G. Genetic heterogeneity of single disseminated tumour cells in minimal residual cancer. Lancet. 2002 Aug 31;360(9334):683-9. doi: 10.1016/S0140-6736(02)09838-0. PMID 12241875
- [Background] Choesmel V, Pierga JY, Nos C, Vincent-Salomon A, Sigal-Zafrani B, Thiery JP, Blin N. Enrichment methods to detect bone marrow micrometastases in breast carcinoma patients: clinical relevance. Breast Cancer Res. 2004;6(5):R556-70. doi: 10.1186/bcr898. Epub 2004 Jul 29. PMID 15318937
- [Derived] Lesurf R, Griffith OL, Griffith M, Hundal J, Trani L, Watson MA, Aft R, Ellis MJ, Ota D, Suman VJ, Meric-Bernstam F, Leitch AM, Boughey JC, Unzeitig G, Buzdar AU, Hunt KK, Mardis ER. Genomic characterization of HER2-positive breast cancer and response to neoadjuvant trastuzumab and chemotherapy-results from the ACOSOG Z1041 (Alliance) trial. Ann Oncol. 2017 May 1;28(5):1070-1077. doi: 10.1093/annonc/mdx048. PMID 28453704
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu